CLINICAL TRIAL: NCT00369226
Title: Phase I/II Trial of Bortezomib (Velcade) in Addition to Tacrolimus and Methotrexate to Prevent Graft Versus Host Disease (GVHD) After Mismatched Allogeneic Non-Myeloablative Peripheral Blood Stem Cell Transplantation
Brief Title: Bortezomib Plus Tacrolimus and Methotrexate to Prevent Graft Versus Host Disease (GVHD) After Mismatched Allogeneic Non-Myeloablative Blood Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, John Koreth, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06-065; X05175
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-06

CONDITIONS: Hematologic Malignancies
Keywords: Velcade; Bortezomib; Allogeneic Stem Cell Transplant; GVHD
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Bortezomib; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib/Tacrolimus/Methotrexate post HSCT (Experimental)
  Interventions: Drug: Bortezomib (Velcade); Drug: Tacrolimus; Drug: Methotrexate; Procedure: blood stem cell transplantation

INTERVENTIONS:
Drug: Bortezomib (Velcade) — Infusion for a total of 3 doses
Drug: Tacrolimus — Taken until Doctor determines it is not necessary any more
Drug: Methotrexate — Infusion for a total of 4 doses
Procedure: blood stem cell transplantation — Allogeneic Non-myeloablative peripheral blood stem cell transplantation

SUMMARY:
The purpose of this study is to determine if Velcade (also known as bortezomib) can help prevent graft versus host disease (GVHD) developing after transplantation. This is done by using a combination of three immune suppressive medications: Velcade, tacrolimus and methotrexate. Stem cell transplantation is one of the options for patients with cancer of the blood or blood forming organs. Recently, allogeneic stem cell transplants have been performed using lower doses of chemotherapy and radiotherapy: non-myeloablative or "mini" transplants. GVHD is a significant problem that may occur even after "mini" transplantations. Information from other research studies, suggests that Velcade may help to reduce the risk of developing GVHD when given early after transplantation.

DETAILED DESCRIPTION:
* In this study we are looking for the highest dose of Velcade that can be given to people safely when given with tacrolimus and methotrexate. Not everyone who participates in the study will receive the same amount of the study drug. The dose the participant will receive depends upon the number of subjects enrolled on the study and how well they have tolerated their doses of the drug.
* Before Transplant: In addition to the chemotherapy drugs, fludarabine and busulfex, for the participants non-myeloablative transplant, they will also start taking tacrolimus orally three days before their transplant.
* After Transplant Medication: Methotrexate; Intravenously on days 1, 3, 6 & 11 after transplant for a total of 4 doses. Tacrolimus; Continue taking orally once daily. Velcade: Intravenously on days 1, 4 & 7 after transplant, a total of 3 doses. Filgrastim: Subcutaneous injection daily starting the day after transplant and continuing until the participant blood counts have recovered.
* After Transplant Physical Exams & Tests: Participants will have physical exams and blood tests every week for 1 month. After 1 month, a none marrow biopsy will be performed to look for evidence of the donor's cells in the participants bone marrow.
* Following the 1 month period of time, participants will be seen every few weeks. Another bone marrow biopsy, as well as blood tests, will be taken 3-4 months after the transplant to review the disease status. At this point, participants will come into the clinic about every 3 months, or as determined by their physician for about one year.
* While the study ends at 12 months after transplant, we would like to keep track of the participants medical condition for the rest of their life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies including myelodysplastic syndrome (MDS), who are at a high risk of complications after myeloablative transplantation
* Patients have a donor (both related and unrelated) who are mismatched according to protocol criteria
* 18 years of age or older
* Performance status 0-2
* Life expectancy of > 100 days
* Female subject is either post-menopausal or sterilized or willing to use an acceptable form of birth control
* Male subject agrees to use an acceptable form of birth control

Exclusion Criteria:

* Evidence of HIV infection
* Total bilirubin > 2.0mg/dl that is due to hepatocellular dysfunction
* Aspartate aminotransferase (AST) > 90
* Known active hepatitis B or C
* Serum creatinine > 2.0
* Greater than or equal to Grade 2 peripheral neuropathy within 21 days of enrollment
* Prior allogeneic stem cell transplant
* Patients with myeloproliferative disease (e.g. myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia)
* Myocardial infarction within 6 months prior to enrollment or has NYHA Class III or IV hear failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Hypersensitivity to Velcade, boron or mannitol
* Pregnant or breast feeding
* Patient has received other investigational drugs 14 days before enrollment
* Serious medical or psychiatric illness
* Another active solid tumor malignancy at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-08; Primary Completion 2010-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, MD, Principal Investigator — Dana-Farber Cance Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Koreth J, Stevenson KE, Kim HT, Garcia M, Ho VT, Armand P, Cutler C, Ritz J, Antin JH, Soiffer RJ, Alyea EP 3rd. Bortezomib, tacrolimus, and methotrexate for prophylaxis of graft-versus-host disease after reduced-intensity conditioning allogeneic stem cell transplantation from HLA-mismatched unrelated donors. Blood. 2009 Oct 29;114(18):3956-9. doi: 10.1182/blood-2009-07-231092. Epub 2009 Aug 27. PMID 19713456

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I (45 Days): Bortezomib plus tacrolimus and methotrexate after mismatched allogeneic non-myeloablative hematopoietic stem cell transplantation (HSCT).
Period: Phase I (45 Days)
Arm/Group | Phase I (45 Days) | Phase II (45 Days)
Started | 13 | 0
Completed | 13 (Once MTD established, additional 10 patients were accrued at MTD to better estimate toxicity.) | 0
Not Completed | 0 | 0
Period: Phase II (45 Days)
Arm/Group | Phase I (45 Days) | Phase II (45 Days)
Started | 0 | 32
Completed | 0 | 32 (This includes 10 patients treated at candidate MTD in Phase I.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 13 | 32 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 25 | 38
  >=65 years | 0 | 7 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 21
  Male | 6 | 18 | 24
Region of Enrollment [Number; unit: participants]
  United States | 13 | 32 | 45

OUTCOME MEASURES:

1. Primary Outcome: The Maximally Tolerated Dose (MTD) of Bortezomib (Velcade) That Can be Administered With Tacrolimus and Methotrexate After Mismatched Allogeneic Non-myeloablative Peripheral Blood Stem Cell (PBSC) Transplantation
Description: The MTD of bortezomib was evaluated at 3 dose levels:
  Dose level 1: 1.0 mg/m^2 Dose level 2: 1.3 mg/m^2 Dose level 3: 1.5 mg/m^2 Cohorts of 3-5 pts were enrolled at each dose level. At any dose level, if no DLT in the first 3, 4, or 5 pts, then dose escalation would occur.
  If 3 evaluable pts in cohort, and 1 of 3 experiences DLT then 2 additional pts treated at the same dose level. If >=1 of 2 additional pts experience DLT then previous dose level will be MTD. If no DLT in additional 2 pts then dose escalation will occur. If 4 evaluable pts in cohort, and 1 of the 4 experiences DLT then 1 additional pt treated at same dose level. If this additional pt experiences DLT then the previous dose will be declared to be the MTD. If additional pt does not experience DLT, then dose escalation will take place. If 5 evaluable pts in cohort, and 1 experiences DLT, then dose escalation will take place. If >=2 of first 3, 4, or 5 pts experience DLT then the previous dose will be declared MTD.
Time Frame: by day 45 post PBSC infusion
Measure: Number; unit: mg/m^2
Arm/Group | Phase I
Number analyzed (Participants) | 13
mg/m^2 | 1.3

2. Primary Outcome: Successful Initial Engraftment by Day 45 Post Peripheral Blood Stem Cell (PBSC) Infusion and Administration of Bortezomib (Velcade), Tacrolimus and Methotrexate
Description: Percentage of participants who did not experience failure to engraft or relapse or death before assessment.
Time Frame: by day 45 post PBSC infusion
Measure: Number; unit: percentage of participants
Groups:
- Combined Phase I Plus Phase II: This reports on the total phase I plus phase II patients who were evaluable for chimerism endpoint (37 of the 45 patients).
Arm/Group | Combined Phase I Plus Phase II
Number analyzed (Participants) | 37
percentage of participants | 97

3. Primary Outcome: Incidence of Grade II-IV Acute Graft Versus Host Disease (GVHD) by Day 100.
Time Frame: by day 100 after peripheral blood stem cell (PBSC) infusion
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase I and Phase II: This reports on all treated patients across both phase I and phase II (n=45)
Arm/Group | Phase I and Phase II
Number analyzed (Participants) | 45
percentage of participants | 22 [11 to 35]

4. Secondary Outcome: Sustained Engraftment Following Transplant.
Description: As measured by median total donor chimerism at day 100.
Time Frame: by day 100 post transplant
Population: Several subjects experienced failure to graft, relapse or death prior to assessment and were removed from analysis.
Measure: Number; unit: percentage of participants
Groups:
- Phase I and Phase II: Engraftment is determined for all treated patients across both phase I and phase II (n=45) who are evaluable for this endpoint (n=35)
Arm/Group | Phase I and Phase II
Number analyzed (Participants) | 35
percentage of participants | 97

5. Secondary Outcome: Incidence of Chronic Graft Versus Host Disease (Chronic GVHD).
Description: Number of participants with chronic GVHD at 1 year post transplant.
Time Frame: by 1 year after PBSC infusion
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I and Phase II
Number analyzed (Participants) | 45
percentage of participants | 29 [16 to 43]

6. Secondary Outcome: Overall Survival and Progression-free Survival.
Description: Progression is defined as disease relapse or disease progression since transplant.
Time Frame: by 1 year after PBSC infusion
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Progression-free Survival (PFS); Overall Survival (OS): This reports on all treated patients across both phase I and phase II (n=45)
Arm/Group | Progression-free Survival (PFS) | Overall Survival (OS)
Number analyzed (Participants) | 45 | 45
percentage of participants | 60 [44 to 73] | 76 [60 to 86]

ADVERSE EVENTS:
Time Frame: By day 45 post PBSC infusion.
Arm/Group | Phase I-II
Serious Adverse Events (participants affected / at risk) | 7/45
Other Adverse Events (participants affected / at risk) | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I-II (N=45)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — CTCAE grade 3
Parainfluenzae sinusitis (Infections and infestations) | 1 (1) — CTCAE grade 3
Cerebrovascular accident with parathesias (Injury, poisoning and procedural complications) | 1 (1) — CTCAE grade 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — CTCAE grade 3
Deep vein thrombosis/pulmonary embolus (Vascular disorders) | 1 (1) — CTCAE grade 3
Clostridium difficile diarrhea (Infections and infestations) | 1 (1) — CTCAE grade 3
Coagulase-negative staphylococcal bacteremia (Infections and infestations) | 1 (1) — CTCAE grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes